CLINICAL TRIAL: NCT06094803
Title: Mindfulness-based Zentangle for Reducing Depression and Anxiety Symptoms in Parents: a Pilot Randomised Controlled Trial
Brief Title: Mindfulness-based Zentangle for Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Grace SUN Yuying, Assistant Professor, Hong Kong Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HE-RD/2023/1.17
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Depressive Symptoms; Anxiety; Well-Being, Psychological
Keywords: Depressive Symptoms; Anxiety; Zentangle; Parents; Mindfulness-based
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receiving Mindfulness-based Zentangle Interventions (Experimental): Participants in the intervention group will receive two 2-hour weekly sessions, focusing on two main themes, which are "Self-awareness and self-kindness" as well as "Acceptance and non-judgmental attitude". Each session with one hour duration and have five different contents separately.
  Interventions: Behavioral: Mindfulness-based Zentangle Program
- Waitlist Control Group (No Intervention): The waitlist control group will not receive any training before all the assessments have been done by both groups. Yet, they will receive the same mindfulness-based Zenatngle training after the assessment period (3 months after baseline). They will be notified that their level of depressive and/or anxiety symptoms when the baseline assessment has been finished. Respondents with Patient Health Questionnaire (PHQ-9) or General Anxiety Disorder (GAD-7) score higher than 14 will be advised to consult a doctor, same as the intervention group.

INTERVENTIONS:
Behavioral: Mindfulness-based Zentangle Program — Session 1 focuses on "Self-awareness and Self-kindness" through the Zentangle method. It covers the introduction, basic techniques, and eight steps of Zentangle. Participants practice mindfulness and learn grid and round patterns. Drawing mindfully and interactive sharing are encouraged for engagement and reflection.
  Session 2 emphasizes "Acceptance and Non-judgmental Attitude". It builds on the previous session, exploring advanced techniques in the Zentangle method. Participants practice mindfulness, learn organic and texturing patterns, create their own artwork, and engage in interactive sharing for reflection.
  Arms: Receiving Mindfulness-based Zentangle Interventions

SUMMARY:
Substantial evidence supports the effect of mindfulness practices on improving health outcomes. Zentangle is a mindfulness-based art therapy (MBAT) that combines art-making and meditation using simple materials. The goal of this pilot randomized controlled trial is to assess the effectiveness of mindfulness-based Zentangle interventions for reducing depression and anxiety symptoms and mindful parenting in parents with mild to severe depression or anxiety. Participants will be instructed to attain the Zentangle courses, a Certified Zentangle Teacher (CZT) will deliver two 2-hour weekly group sessions. At the end of the course, they will be invited to participate in an artwork show. After completing the assessments, the waitlist control group will receive the same training sessions and also be invited to the artwork show. The hypothesis is that the intervention group will show more significant decreases in depressive and anxiety symptoms, mental well-being and mindful parenting improvement, less stress and better quality of life than the control group.

DETAILED DESCRIPTION:
Parents face day-to-day stress related to parenting and other stressors, such as low household income, child behavioural problems and high expectations for their children. Mindful parenting research is becoming popular in recent years, and substantial evidence supports the effect of mindfulness practices on improving health outcomes. The simplicity of Zentangle gives it the potential to cultivate and apply mindfulness practice in daily family life. Zentangle art is becoming popular in Hong Kong and in other countries and regions. However, there are limited exploratory trials to evaluate the effectiveness of Zentangle. Therefore, the aim of the present study is to assess the effectiveness of mindfulness-based Zentangle interventions for reducing depression and anxiety symptoms in parents with mild to moderate depression or anxiety.

A pilot randomised controlled trial (1:1 allocation ratio) on parents who have mild to severe depression or anxiety symptoms will be conducted. Participants will be approached through public posters or active approach in community centres, such as Caritas Community Centre. Interested individuals will scan the QR code on the poster and complete a short online questionnaire via Qualtrics. The research staff will contact the eligible respondents and send them a link for collecting the baseline questionnaire (T1). Randomisation will be conducted after obtaining consent and completion of T1. Participants will be randomised into the intervention or control groups using random numbers generated by a statistician not involved in any part of the study. The random numbers will be generated by Microsoft Excel. The recruitment staff will be concealed from the allocation process. The intervention group will receive two weekly sessions of training and complete the immediate post-intervention assessment (T2, two weeks after T1), and the 3-month assessment (T3, three months after T1). The waitlist control group will complete the assessments during the same time points and receive the training after completion of T3.

A Certified Zentangle Teacher (CZT) will deliver two 2-hour weekly group sessions to the intervention group. The content will include 1) an introduction to Zentangle, guide participants to set intentions of mindfulness, open mind, gratitude, and appreciation; 2) simple mindfulness practice in each session to cultivate mindfulness, such as body scan and sitting meditation; 3) step-by-step explanation and demonstration of examples of various patterns; 4) instruct participants to create their unique art; 5) interactive sharing of participants' artworks, experience and feelings during the workshop. After completing the assessments, the waitlist control group will receive the same training sessions. An art show will be organised afterwards. Parents will be invited to create one or two pieces of Zentangle artwork at home and submit them to the research team before the show.

The baseline characteristics of the two groups will be compared using an independent t-test and Chi-squared test. An intention-to-treat approach will be used and a multilevel mixed model will be built to calculate between-group mean differences in the outcomes after adjusting for the baseline values of the respective outcomes. The effect size (Cohen's d) will be calculated. Subgroup analyses will also be conducted based on the number of drawings actually performed by participants. Within-group mean differences will be compared by paired t-tests. Missing data were recognised as randomly missing and dealt with the multiple imputation method. A complete case analyses will performed as a sensitivity analysis. It is expected that the intervention group show more significant improvements in the measured outcomes than the control group, indicating preliminary evidence of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Parents with children in primary or secondary schools (Grade P1-6 and S1-6, 6-17 years old), being between 24 and 59 years old;
2. Report mild to severe depressive symptoms (score of 5-27 on the Patient Health Questionnaire, PHQ-9) or anxiety (General Anxiety Disorder (GAD) - 7, score 5-21) during the screening. Respondents with PHQ or GAD score > 14 will be advised to consult a doctor.
3. Hong Kong residents who can speak Cantonese and read Chinese;
4. Individuals who have interests in participation and are able to communicate.

Exclusion Criteria:

1) under psychiatric treatment or taking antidepressants in the past six months;

Ages: 24 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in Depressive Symptoms | T1: Baseline; T2: Immediate post-intervention; T3: Three months after the intervention
  Depressive symptoms will be assessed using the Patient Health Questionnaire (PHQ)-9. Participants will be asked to rate the frequency of nine symptoms experienced in the past two weeks on a 4-point Likert scale, ranging from 0 (not at all) to 3 (nearly every day). The total score on the PHQ-9 ranges from 0 to 27, with higher scores indicating a higher severity of depressive symptoms.
Changes in Anxiety Symptoms | T1: Baseline; T2: Immediate post-intervention; T3: Three months after the intervention
  To assess anxiety disorder, the Generalized Anxiety Disorder (GAD)-7 scale will be adopted. Participants will rate the frequency of seven symptoms on a 4-point Likert scale (from 0=not at all to 3=nearly every day), using the same response options as the PHQ-9 scale. The total score on the GAD-7 ranges from 0 to 21, with a higher score indicating a greater level of anxiety.

SECONDARY OUTCOMES:
Changes in Well-being | T1: Baseline; T2: Immediate post-intervention; T3: Three months after the intervention
  The Short Warwick-Edinburgh Mental Well-being Scale, consisting of seven items, will be utilized to assess well-being. Participants will use a 5-point Likert scale (1=none of the time, 5=all the time) to rate their experiences. The well-being score is determined by summing the responses to all seven items, resulting in a range of 7 to 35. A higher score indicates a greater level of well-being.
Changes in Perceived Psychological Stress | T1: Baseline; T2: Immediate post-intervention; T3: Three months after the intervention
  To assess psychological stress over the past month, the Chinese version of the Perceived Stress Scale-10 (PSS-10) will be employed. The scale comprises six positive and four negative items, with each item rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The positive items will be reverse scored before calculating the total score. Scores on the PSS-10 range from 0 to 40, with higher scores indicating a greater perceived psychological stress level.
Quality-adjusted Life Years (QALYs) | T1: Baseline; T2: Immediate post-intervention; T3: Three months after the intervention
  The 5-item EuroQol (EQ-5D-5L) will be used to measure the QALYs. The crosswalk value sets of Hong Kong will be used to convert EQ-5D-5L to the utility weight. The values ranged from -0.864 to 1. Each individual QALY was calculated by using the Area Under the Curve method.
Mindfulness in Parenting | T1: Baseline; T2: Immediate post-intervention; T3: Three months after the intervention
  To evaluate mindful parenting for parents with children or/and adolescents, ranging in age from 2 to 16 years old, the Chinese version of the Mindfulness in Parenting Questionnaire (MIPQ) will be used. Participants will use a 4-point Likert scale (1=sometimes, 4=all the time) to rate their experiences. The score is determined by summing the responses to all 28 items, resulting in a range of 28 to 112. A higher score indicates a higher level of mindful parenting.

OTHER OUTCOMES:
Overall satisfaction with the program and subjective changes | T2: Immediate post-intervention; T3: Three months after the intervention
  Subjective changes including personal mental health, parent-child conflict, and parent-child communication. Participants will rate their overall satisfaction with the activity on a scale of 0 to 10, where "0" represents "very unsatisfied" and "10" represents "very satisfied". Open-ended questions will be used to gather comments and suggestions from the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Yuying Sun, Principal Investigator — Hong Kong Metropolitan University
Locations (1):
- Jockey Club Institute of Healthcare, Hong Kong Metropolitan University, Hong Kong, Hong Kong